CLINICAL TRIAL: NCT07284004
Title: Metabolic Dysfunction Associated Fatty Liver Disease in Long-Term Cholecystectomy Patiens
Brief Title: Fatty Liver in Long Standing Cholecystectomy
Acronym: MAFLD-Chole St
Status: Not yet recruiting | Type: Observational
Sponsor: Yasmeen Ahmed Farrag Ahmed (Other)
Responsible Party: Sponsor-Investigator, Yasmeen Ahmed Farrag Ahmed, Resident Doctor Tropical Medicine and Gastroenterology, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med--25-11-6MS
Record Dates: First submitted 2025-11-30; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD)-Post-cholecystectomy Metabolic Changes -Hepatic Steatosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Long-term cholecystectomy patients

SUMMARY:
This observational study aims to evaluate the association between long-term cholecystectomy and the development of metabolic dysfunction-associated fatty liver disease (MAFLD) in adult patients. The study will assess the prevalence and severity of hepatic steatosis in individuals who underwent cholecystectomy several years earlier and compare clinical, metabolic, and biochemical parameters to identify potential risk factors. The goal is to determine whether cholecystectomy contributes to metabolic alterations that increase the likelihood of MAFLD in the long term.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

1. Patients less than 18 years old.
2. Body mass index (BMI) ≤ 25 kg/m2
3. Patients with chronic renal failure.
4. Patients with liver cirrhosis.
5. Patients with acute liver dysfunction.
6. Breast feeding and pregnancy.
7. patients have done cholecystectomy less than 5 years ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) who have undergone cholecystectomy at least 5 years prior to enrollment, with no known chronic liver diseases other than metabolic dysfunction-associated fatty liver disease (MAFLD). Participants will be recruited from outpatient gastroenterology clinics and will provide informed consent before enrollment. Both male and female patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of metabolic dysfunction-associated fatty liver disease (MAFLD) in patients after long term follow up post cholecystectomy | 5 years post-cholecystectomy

SECONDARY OUTCOMES:
Changes in serum level of ALT in post-cholecystectomy patients | Annually for 5 years

IPD SHARING:
Plan to Share IPD: Undecided